CLINICAL TRIAL: NCT02817451
Title: Immunogenicity and Safety of Sanofi Pasteur's DTaP-IPV-HB-PRP-T Combined Vaccine Given as a Primary Series and a Second Year of Life Booster in HIV-Exposed Infected and in HIV-Exposed Uninfected Infants in Republic of South Africa
Brief Title: DTaP-IPV-HB-PRP-T Combined Vaccine as a Primary Series and a Second Year of Life Booster in HIV-Exposed Infected and Uninfected Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L44; U1111-1161-2610 (Other: WHO); 2018-004708-21 (EudraCT Number)
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Polio; Human Immunodeficiency Virus Infection
Keywords: Diphtheria; Tetanus; Pertussis; Hepatitis B; DTaP IPV HB PRP-T Combined Vaccine; Human Immunodeficiency Virus
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Acquired Immunodeficiency Syndrome | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group A (Experimental): HIV exposed and infected infants
  Interventions: Biological: Hexaxim®: DTaP-IPV-HB-PRP-T Combined Vaccine
- Study Group B (Experimental): HIV exposed and uninfected infants
  Interventions: Biological: Hexaxim®: DTaP-IPV-HB-PRP-T Combined Vaccine

INTERVENTIONS:
Biological: Hexaxim®: DTaP-IPV-HB-PRP-T Combined Vaccine — 0.5 mL, Intramuscular at 6, 10, and 14 weeks of age + a booster at age 15 to 18 months
  Other Names: Hexaxim®
  Arms: Study Group A
Biological: Hexaxim®: DTaP-IPV-HB-PRP-T Combined Vaccine — 0.5 mL, Intramuscular at 6, 10, and 14 weeks of age + a booster at age 15 to 18 months
  Other Names: Hexaxim®
  Arms: Study Group B

SUMMARY:
This study aims to assess and confirm the adequate immunogenicity and safety profile of the Sanofi Pasteur's DTaP-Hep B-IPV-PRP-T fully liquid combined hexavalent vaccine administered in HIV-exposed uninfected infants and in HIV-exposed infected infants.

The primary objectives of the study are:

* To evaluate the immunogenicity of the study vaccine 1 month after the 3-dose primary series in HIV-exposed infected and in HIV-exposed uninfected infants.
* To describe the persistence of all antibodies before receipt of the booster dose in HIV-exposed infected and in HIV-exposed uninfected infants.
* To evaluate the immunogenicity of the study vaccine 1 month after the booster dose in HIV-exposed infected and in HIV-exposed uninfected infants.

The secondary objectives of the study are:

* To describe the safety profile after each and all doses of the study vaccine administered as a 3-dose infant primary series in HIV-exposed infected and in HIV-exposed uninfected infants.
* To describe the safety profile of the study vaccine administered as a booster in HIV-exposed infected and in HIV-exposed uninfected infants.

DETAILED DESCRIPTION:
Male and female infants born from HIV-infected mothers will be tested for HIV infection from birth to 6 weeks of age. HIV infected and HIV uninfected participants will be enrolled into two groups at Day 0. Some infants detected HIV-exposed infected outside of the hospital center facilities and the trial screening procedure may also be enrolled. All participants will receive primary vaccinations with Sanofi Pasteur's DTaP-IPV-HB-PRP-T combined vaccine at 6, 10 and 14 weeks of age and a booster dose at approximately 15 to 18 months of age will receive a booster dose of the Sanofi Pasteur's DTaP-IPV-HB-PRP-T combined vaccine.

ELIGIBILITY:
Inclusion Criteria:

(Screening Criteria for the participants mother)

* At least 18 years of age at the time of the Screening blood sample draw
* Self-reported or maternity-reported HIV infection in the mother

Inclusion Criteria:

* Born to an adult mother and aged 35 to 56 days (between 5 and 8 weeks of age) on the day of inclusion
* Group A participants must be HIV infected, as documented through the results of a polymerase chain reaction (PCR) test, and following an anti-retroviral therapy according to the national recommendations; and Group B participants must be HIV exposed uninfected infants, as documented through the results of a PCR test.
* Born with a birth weight ≥ 2.0 kg
* Informed consent form signed by the parent(s)/legal guardian(s) and by one independent witness if the parent(s)/legal guardian(s) is illiterate
* Participants and parent(s)/legal guardian(s) are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial of an investigational product in the 4 weeks preceding the trial inclusion (receipt of study vaccine) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Group A participants diagnosed with a chronic condition, except HIV infection, or any experience of blood or blood-derived products received or experience of thrombocytopenia or bleeding disorder; and Group B participants diagnosed with chronic illness or any experience of blood or blood-derived products received or experience of thrombocytopenia or bleeding disorder.
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis (oral polio vaccine [OPV] given at birth does not constitute an exclusion criteria), hepatitis B (a birth dose of Hep B vaccine does not constitute an exclusion criteria) diseases or Hib infection with the trial vaccine or another vaccine. Previous vaccination with Bacillus Calmette-Guerin (BCG) is not considered an exclusion criterion
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, or Haemophilus influenzae type b infections (confirmed either clinically, serologically or microbiologically)
* History of seizures or history of uncontrolled neurologic disorder or uncontrolled epilepsy until treatment for the condition has been established, the condition has stabilized and the benefit clearly outweighs the risk
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Febrile (axillary temperature ≥ 38°C) or acute illness on the day of inclusion (temporary contraindication).

Ages: 5 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Anti-Pertussis Toxoid (PT) and Anti-Filamentous Hemagglutinin (FHA) Antibody (Ab) Concentrations >= Lower Limit of Quantification (LLOQ) and >=4*LLOQ at Baseline | Day 0 (baseline)
  Anti-PT and anti-FHA Ab concentrations are determined in terms of endotoxin units per millilitre (EU/mL).
Geometric Means of Anti-Pertussis Toxoid and Anti-Filamentous Hemagglutinin Antibody Concentrations at Baseline | Day 0 (baseline)
  Anti-PT and anti-FHA Ab levels are measured by electrochemiluminescence immunoassay (ECL) and anti-PT and anti-FHA Ab concentrations are determined in terms of EU/mL.
Geometric Means of Antibody Titers/Concentrations After Primary Series Vaccination | Day 90 (1 month after third dose)
  Anti-diphtheria, anti-tetanus, anti-PT and anti-FHA Ab levels are measured by ECL. Anti-poliovirus types 1, 2, and 3 Ab levels are measured by neutralisation assay. Anti-Hep B Ab levels are measured by VITROS ECi/ECiQ Immunodiagnostic system using chemiluminescence detection technology. Anti-polyribosylribitol phosphate (PRP) Ab levels are measured using a Farr-type radioimmunoassay (RIA). Ab concentrations are determined as: anti-diphtheria >=0.01 international units (IU)/mL, >=0.1 IU/mL, 1.0 IU/mL, anti-tetanus >=0.01 IU/mL, >=0.1 IU/mL, and >=1.0 IU/mL, anti-PT and anti-FHA EU/mL, anti-PRP >=0.15 microgram (mcg)/mL, >=1.0 mcg/mL, anti-Poliovirus types 1, 2, and 3 Ab titers >=8 (1/dilution [dil]), Anti-Hep B >=10 milli (m) IU/mL, and >=100 mIU/mL.
Number of Participants With Seroprotection After Primary Series Vaccination | Day 90 (1 month after third dose)
  Seroprotection is determined as: anti-diptheria Ab concentrations >=0.01 IU/mL, >=0.1 IU/mL, and >=1.0 IU/mL, anti-tetanus Ab concentrations >=0.01 IU/mL, >=0.1 IU/mL, and >=1.0 IU/mL, anti-PT and anti-FHA Ab concentrations EU/mL (>=LLOQ and >=4*LLOQ), anti-PRP Ab concentrations >=0.15 mcg/mL and >=1.0 mcg/mL, anti-poliovirus 1, 2, and 3 Ab titers >=8 (1/dil), anti-Hep B Ab concentrations >=10 mIU/mL and >=100 mIU/mL.
Number of Participants with Vaccine Response or Seroconversion After Primary Series Vaccination | Day 0 (baseline), Day 90 (1 month after third dose)
  Vaccine response is defined for anti-PT and anti-FHA as Ab post-Dose 3 concentrations >=4*LLOQ, if pre-Dose (Day 0) Ab concentration is <4*LLOQ or 1 month after third dose (Day 90) concentrations >= pre-Dose Ab concentrations if pre-Dose (Day 0) concentrations >=4*LLOQ. Seroconversion for anti-PT and anti-FHA is defined as >=4-fold Ab concentrations increase from pre-Dose (Day 0) to 1 month after third dose (Day 90).
Geometric Means of Antibody Titers/Concentrations After Booster Vaccination | Day 420 (1 month after booster vaccination)
  Anti-diphtheria, anti-tetanus, anti-PT, and anti-FHA Ab levels are measured by ECL. Anti-poliovirus types 1, 2, and 3 Ab levels are measured by neutralisation assay. Anti-Hep B Ab levels are measured by VITROS ECi/ECiQ Immunodiagnostic system using chemiluminescence detection technology. Anti-PRP Ab levels are measured using a Farr-type RIA. Ab concentrations: anti-diphtheria >=0.01 IU/mL, >=0.1 IU/mL, >=1.0 IU/mL, anti-tetanus >=0.01 IU/mL, >=0.1 IU/mL, and >=1.0 IU/mL, anti-PT and anti-FHA EU/mL, anti-PRP >=0.15 mcg/mL, >=1.0 mcg/mL, anti-poliovirus 1, 2, and 3 Ab titers >=8 (1/dil), anti-Hep B >=10 mIU/mL, and >=100 mIU/mL.
Number of Participants With Seroprotection After Booster Vaccination | Day 420 (1 month after booster vaccination)
  Seroprotection: anti-diphtheria Ab concentrations >=0.01 IU/mL, >=0.1 IU/mL, and >=1.0 IU/mL, anti-tetanus Ab concentrations >=0.01 IU/mL, >=0.1 IU/mL, and >=1.0 IU/mL, anti-PT and anti-FHA Ab concentrations EU/mL (>=LLOQ and >=4*LLOQ), anti-PRP Ab concentrations >=0.15 mcg/mL and >=1.0 mcg/mL, anti-poliovirus 1, 2, and 3 Ab titers >=8 (1/dil), and anti-Hep B Ab concentrations >=10 mIU/mL and >=100 mIU/mL.
Number of Participants With Vaccine Response or Seroconversion After Booster Vaccination | Day 0 (baseline), Day 420 (1 month after booster vaccination)
  Vaccine response is defined for anti-PT and anti-FHA as >=4 fold Ab concentrations increase from pre-dose (Day 0) to 1 month after booster dose (Day 420), if pre-Dose (Day 0) Ab concentrations <4*LLOQ; or >=2 fold Ab concentrations increase from pre- dose (Day 0) to 1 month after booster dose (Day 420), if pre-dose (Day 0) Ab concentrations >=4*LLOQ. Seroconversion is defined for anti-PT and anti-FHA as >=4 fold Ab concentrations increase from pre-dose (Day 0) to 1 month after booster dose.
Number of Participants With Booster Response After Booster Vaccination | Day 390 (pre-booster), Day 420 (1 month after booster dose)
  Booster response is defined for anti-PT and anti-FHA as >=4 fold Ab concentrations increase from pre-booster (Day 390) to 1 month after booster dose (Day 420), if pre-booster Ab concentrations <4*LLOQ; or >=2 fold Ab concentrations increase from pre-booster (Day 390) to 1 month after booster dose (Day 390) if pre-Booster Ab concentrations >=4*LLOQ.

SECONDARY OUTCOMES:
Number of Participants With Immediate Unsolicited Adverse Events (AE) After Primary Series Vaccination | Within 30 minutes after vaccination
  An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the electronic case report form (eCRF) in terms of diagnosis and/or onset post-vaccination.
Number of Participants With Solicited Injections Site or Systemic Reactions After Primary Series Vaccination | Within 7 days after vaccination
  A solicited reaction is an adverse reaction observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited injection site reactions: injection site tenderness, erythema, and swelling. Solicited systemic reactions: fever, vomiting, crying abnormal, drowsiness, appetite lost, and irritability
Number of Participants With Unsolicited Adverse Events After Primary Series Vaccination | Within 30 days after vaccination
  An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of diagnosis and/or onset post-vaccination. An unsolicited non-serious AE is an unsolicited AE excluding serious adverse events (SAEs). Systemic AEs are all AEs that are not injection site reactions. They therefore include systemic manifestations such as headache, fever, as well as localized or topical manifestations that are not associated with the vaccination site.
Number of Participants With Serious Adverse Events During the Study | Day 0 to Day 420
  An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event.
Number of Participants With Immediate Unsolicited Adverse Events After Booster Vaccination | Within 30 minutes after booster vaccination
  An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of diagnosis and/or onset post-vaccination.
Number of Participants With Solicited Injection Site or Systemic Reactions After Booster Vaccination | Within 7 days after booster vaccination
  A solicited reaction is an adverse reaction observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited injection site reactions: tenderness, erythema, swelling, and extensive limb swelling. Solicited systemic reactions: fever, vomiting, crying abnormal, drowsiness, appetite lost, and irritability.
Number of Participants With Unsolicited Adverse Events After Booster Vaccination | Within 30 days after booster vaccination
  An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of diagnosis and/or onset post-vaccination. An unsolicited non-serious AE is an unsolicited AE excluding SAEs. Systemic AEs are all AEs that are not injection site reactions. They therefore include systemic manifestations such as headache, fever, as well as localized or topical manifestations that are not associated with the vaccination site.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur SA
Locations (1):
- Soweto, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org